CLINICAL TRIAL: NCT07179497
Title: Evaluation of the Safety and Performance of the Neobone®: A Prospective Observational Study in Dental Area
Acronym: NeoDent01
Status: Recruiting | Type: Observational
Sponsor: Bioceramed (Industry)
Collaborators: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Responsible Party: Sponsor
Other Study IDs: NeoDent01
Record Dates: First submitted 2025-09-05; First posted 2025-09-17 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Bone Augmentation
Keywords: prospective observational clinical study; bone substitute; bone defects; hydroxyapatite and beta tricalcium phosphate; Neobone®; real-world clinical data; safety; performance; medical device; reconstructive dental surgeries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to collect real-world clinical data to gather information on the performance and safety of the Neobone® when used according to its intended purpose and current clinical applications. The results of the clinical study will serve as clinical evidence for the device's clinical evaluation.

DETAILED DESCRIPTION:
Neobone® is a synthetic and resorbable implantable synthetic calcium phosphate ceramic bone substitute, composed of hydroxyapatite and beta-tricalcium phosphate. The structures composed of these calcium phosphate ceramic structures are rapidly osseointegrated due to its chemical composition, which is similar to the mineral phase of the human bone, and due to the interconnected porosity allowing a total vascularization of the implant. Since beta-tricalcium phosphate is more soluble than hydroxyapatite, this biphasic composition enhances the ceramic resorption, allowing a resorption rate compatible with the physiology of bone cells. Neobone® is a single use, gamma radiation sterilized medical device.

Neobone® is a single use, gamma sterilized, implantable biodegradable medical device intended to be used in filling bony voids or gaps within the skeletal system that do not contribute to the structural stability of the bone, and in reconstructive dental and maxillofacial surgeries. These defects may arise from surgical procedures or result from osseous damage due to traumatic injury to the bone.

Neobone® is intended to be used in operating rooms by trained orthopaedic surgeons, as well as in dental offices or operating rooms by dentists and maxillofacial surgeons who have medical and technical knowledge in bone grafting. Neobone® is a class III medical device and is intended for long-term use and will be placed in contact with cancellous tissue and adjacent tissues through surgically invasive techniques.

This observational post-market study will collect data relating to standard practice procedures, therefore there are no additional risks or direct benefits associated with participating in this registry for the patient.

Participation in the study may provide a better understanding of treatment with Neobone® and potentially influence future clinical decisions, contributing to the continuous improvement of healthcare.

This study based on observations of clinical practice aims to collect clinical data to keep up to date the information on the performance and safety of the medical device when used in accordance with its intended use and current clinical applications. The results of the clinical study shall be used as clinical evidence for clinical evaluation of the medical.

The post-market study is meant to identify and analyse emerging risks, ensure the continued acceptability of the benefit/risk ratio and also identify possible systematic misuse or unauthorized use of the medical device. This protocol does not include any planned new uses, new populations, new materials or design changes.

The results from the prospective observational post-market study will provide clinical evidence on the device's performance and safety in the post-market phase.. This complements the data collected during the pre-market phases, thus protecting patient safety. Active surveillance of the safety of medical devices, achieved through the continuous monitoring of vast sources of clinical data, is a priority in the field of medical devices, a requirement of MDR - Medical Device Regulation No. 2017/745. This approach is crucial to achieving the objectives set, guaranteeing the safety and efficacy of the devices in circulation.

The clinical study population consists of adult patients (aged > 18 years old) who undergo reconstructive dental surgery using the Neobone® medical device. Patients will be followed as per local standard medical practices of the centre for 2 years. Clinical data will be collected at 6 points in time: Visit 1 (before surgery - baseline and enrolment), Visit 2 (moment after surgery), Visit 3 (7 ± 1 days), Visit 4 (6 months ±3 weeks), Visit 5 (12 months ±30 days) and Visit 6 (23 months ±30 days).

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females (age > 18 years old);
* Patients who are able to sign an informed consent form (for data collection);
* Patients undergoing reconstructive dental surgery and indicated for the use of Neobone®;

Exclusion Criteria:

* Patients who are unable to understand consent and the objectives of the study;
* Signs of local or systemic acute/ active or chronic infections;
* Metabolic affections;
* Severe degenerative diseases, conditions in which general bone grafting is not advisable;
* Implementation sites that allow product migration;
* Conditions which require structural support in the skeletal system;
* Conditions where the implantation site is unstable and not rigidly fixated;
* Sensibility to the implantable materials;
* Known hypersensitivity to the implant material.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The clinical study population consists of adult patients (aged > 18 years old) who undergo reconstructive dental surgery using the Neobone® medical device.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Clinical and radiographic performance endpoint: | 6 months
  - Bone gain (augmentation volume in mm³) at 6 months, assessed by computed tomography (CBCT);
Safety Endpoint | Visit 2 (moment after surgery), Visit 3 (7 ± 1 days), Visit 4 (6 months ±3 weeks), Visit 5 (12 months ±30 days) and Visit 6 (23 months ±30 days).
  The assessment of adverse events (AE) and device deficiencies (DD) during the patient follow-up period relation to the medical device. This endpoint will be evaluated at each follow-up visit.
Clinical and radiographic performance endpoint: | 6 months
  - Bone regeneration at the surgical site, clinically viable for implant placement at 6 months (Yes/No), defined as sufficient bone volume and quality, based on clinical evaluation and CBCT, allowing safe implant placement;

SECONDARY OUTCOMES:
Technical success rate | moment after surgery
  Technical success rate and surgeon's satisfaction with the medical device, assessed through a post-surgical questionnaire evaluating usability and overall performance.
Quality of life assessment | Visit 1 (before surgery - baseline and enrolment), Visit 2 (moment after surgery), Visit 3 (7 ± 1 days), Visit 4 (6 months ±3 weeks), Visit 5 (12 months ±30 days) and Visit 6 (23 months ±30 days).
  Quality of life will be assessed using the Oral Health Impact Profile (OHIP-14) questionnaire, administered at baseline, immediately post-surgery, and within the first 7 days postoperatively and during follow-up visits at 6, 12, and 23 months.
Radiographic bone density assessment | 6 months
  Radiographic bone density (Hounsfield units) at 6 months, assessed by CBCT in the regenerated area. The grayscale values (or relative density measurements) will be used to estimate the degree of bone mineralization in the treated site. Elevated radiographic bone density values indicate good mineralization and quality of the regenerated bone. These data serve as complementary indicators of the quality of the bone tissue obtained with the use of the synthetic bone substitute.
Pain level assessment | Visit 1 (before surgery - baseline and enrolment), Visit 2 (moment after surgery), Visit 3 (7 ± 1 days), Visit 4 (6 months ±3 weeks), Visit 5 (12 months ±30 days) and Visit 6 (23 months ±30 days).
  Pain level will be reported using the Visual Analogue Scale (VAS, 0-10), assessed at baseline, immediately post-surgery, within the first 7 days post-operatively, and during follow-up visits at 6, 12, and 23 months.
Bone volume variation (in %) assessment | 6 months
  Bone volume variation (in %) assessed using scans taken at baseline and at 6 months. Volumetric analysis will be performed by superimposing two CBCT images, with the system automatically calculating the percentage difference. This allows quantification of bone gain or maintenance over time. Positive values indicate bone gain, zero indicates maintenance of bone volume, and negative values indicate bone loss. A greater positive volume variation indicates more effective bone regeneration, reflecting a successful outcome at the treated site.

CONTACTS AND LOCATIONS:
Overall Officials: João Botelho, Principal Investigator — Egas Moniz School of Health and Science Caparica
Locations (1):
- Egas Moniz School of Health and Science Caparica, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No